CLINICAL TRIAL: NCT01508546
Title: Conservative Surgery With or Without Axillary Lymphnode Removal in Treating Women With T1N0 Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Roberto Agresti, MD, Principal investigator, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/98
Record Dates: First submitted 2011-12-15; First posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Female Breast Neoplasms; Carcinoma, Ductal, Breast
Keywords: breast cancer; axillary dissection
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: breast surgery with axillary lymphnodes removal (Experimental)
  Interventions: Procedure: axillary dissection
- Arm 2: breast surgery without axillary lymphnodes removal (Experimental)
  Interventions: Procedure: axillary dissection

INTERVENTIONS:
Procedure: axillary dissection — Conservative breast surgery with or without axillary dissection

SUMMARY:
Rationale

Axillary surgery is still fundamental part of breast cancer (BC) management for adjuvant treatment planning.

Purpose

Randomized phase III trial to compare the effectiveness of surgical therapy with or without axillary dissection following conservative treatment in women with stage I breast cancer.

To determine the possibility to avoid axillary surgery in patients with early breast cancer, finding an alternative method to define the need of adjuvant treatment without compromising long-term disease control.

DETAILED DESCRIPTION:
OBJECTIVES:

To compare the efficacy of conservative surgery, with or without axillary lymphnode removal (quadrantectomy with axillary dissection (QUAD) vs. quadrantectomy alone (QU)) followed by adjuvant treatment.

To plan no adjuvant therapy vs. adjuvant therapy (eA+CMF+TAM regimen) based on a biological panel of the primary tumor in the QU group (defined as good panel (GP) ( ER+, and up to one unfavourable features (G3, Her2+++, Laminin Receptor+) or bad panel (BP)(ER-, or ER+ and more than one unfavourable features), whereas in QUAD group based on good factor ( N-, ER+ and GI-II disease (GF)) or bad factor ( N+ or GIII or ER- disease (BF)).

To determine the relationship between the biological variables (hormone receptor status, grading, Laminin receptor, and c-erbB2) and the clinical outcome of the disease in these patients.

OUTLINE This is a randomized unicenter study. Patients are randomized to 1 o 2 treatment arms.

Arm 1: patients undergo conservative surgery with axillary lymphnodes removal Arm 2: patients undergo conservative surgery without axillary lymphnodes removal Post-operative adjuvant strategy was previously described.

Patients are followed every 4 months for the first two years, every 6 months for the following two years, and then annually thereafter.

PROJECT ACCRUAL 600 patients will be accrued for this study over 4 years

ELIGIBILITY Ages eligible for study: 18-65 years Genders eligible for study: female

ELIGIBILITY:
Inclusion Criteria:

* women with T1N0M0 invasive breast cancer
* 18-65 years

Exclusion Criteria:

* bilateral breast cancer
* no other prior or concurrent malignancy except basal cell carcinoma

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 1998-05; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Difference in breast cancer mortality and overall survival between the two arms | median follow-up time: 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Agresti, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- [Derived] Agresti R, Sandri M, Capri G, Bianchi G, Triulzi T, Lozza L, Trecate G, Trapani A, Ferraris C, Paolini B, Menard S, Greco M, Folli S, Tagliabue E. Axillary surgery versus no-axillary staging in T1N0 breast cancer: 20-year follow-up of the INT 09/98 randomized clinical trial. Br J Surg. 2025 Mar 4;112(3):znae311. doi: 10.1093/bjs/znae311. PMID 40042985